CLINICAL TRIAL: NCT00437736
Title: Phase I Dose Finding and Pharmacokinetic Study of Intravenous APO010, a Recombinant Form of Human Fas Ligand, in Patients With Solid Tumors
Brief Title: A Phase I Dose Finding Study of APO010 in Patients With Solid Tumors
Acronym: AP1001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP1001; S065APO01
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Cancer
Keywords: solid tumor; phase I study; dose-escalation
MeSH Terms: conditions — Neoplasms | interventions — Mega-Fas-ligand

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm dose escalation (Experimental)
  Interventions: Drug: APO010

INTERVENTIONS:
Drug: APO010 — APO010 starting at 2.5 µg/m² IV on D1, D15, D22 and D29 followed by a two-week drug rest.

SUMMARY:
Two-centre, open label, uncontrolled, dose-finding phase I study, to determine the safety and tolerability of APO010 administered by intravenous bolus injection once per week. It will be the first time this agent will be administered to humans. At lower dose levels, the first cycle duration is 7 weeks. In subsequent cycles, APO010 is administered as 4 weekly doses followed by a two-week drug rest, cycle duration is 6 weeks. Based on preclinical studies of APO010 may cause liver toxicity and a drop in platelets, that recover within 5 days. The main aim of the study is to identify the recommended dose of APO010 for future clinical studies of APO010.

DETAILED DESCRIPTION:
Two-centre, open label, uncontrolled, dose-finding phase I study, to determine the safety and tolerability of APO010 administered by intravenous bolus injection once per week in patients with solid tumors, for whom therapy of proven efficacy does not exist or is no longer effective. The dose-escalations will follow a classical Fibonacci schedule, meaning at least three patient per dose-level, prior to further escalation. The dose-level assignment and patient registration is centralized by SENDO-Switzerland & Milan offices.

APO010, Apoxis' proprietary humanized recombinant mega-Fas-ligand, is a novel "First in class" investigational anticancer agent. APO010 is a protein that by specific binding to its cognate Fas receptor on the cell surface induces apoptosis (programmed cell death). This is called the extrinsic apoptotic pathway of cells. APO010 has shown to exert anticancer activity in vitro and in animal models carrying a human xenograft of a variety of cancers, including malignancies such as multiple myeloma, non-small cell lung cancer (NSCLC), ovarian cancer. Its activity is cell cycle independent, it does not cross react with known multi-drug resistance mechanism (MDR) and appears to be synergistic with a variety of commonly used anticancer drugs. Hence, APO010 may an attractive candidate for combination anticancer therapy and may be a effective drug in overcoming MDR.

In this study the starting dose is 2.5 microgram/m2. Normally 1/6 of the No-observed-adverse-effect level (NOAEL) dose-level in monkeys would be chosen as the first dose-level, however it has been decided to start at 25% of that dose-level. Across species (mice, rats and Cynomolgus monkeys) the rise in transaminases and drop in platelets occurred at 30 microgram/m2. The Nadir of these toxicities occurred within 6 hours and full recovery at day 5 after the bolus injection.

At the first occurrence of non-reversible (within 1 week) Common Toxicity Criteria (CTC) v3.0 Grade 2 liver function toxicity (Aspartate transaminase (AST)/Alanine transaminase (ALT) or alkaline phosphatase), i.e. Dose Limiting Toxicity (DLT), the patient accrual will be placed on hold until recovery and the subsequent timing of patient accrual to the existing and subsequent cohorts will be re-defined by the sponsor, the principal investigators and SENDO.

Pharmacokinetic assessments will be carried out in all patients during the first, and in consenting patients during the second cycles of treatment.

Assessment for immunogenicity (binding and/or neutralizing antibodies against APO010 will be carried out in all patients in all cycles of treatment before each dose and 2 weeks after the final dose.

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological diagnosis of non-resectable solid tumors for which therapy of proven efficacy does not exist or is no longer effective.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
* Ongoing toxicity associated with prior anticancer therapy ≤Grade 1 (NCI-CTCAE v.3.0).
* No more than 3 prior chemotherapy lines for advanced disease (not including neo/adjuvant chemotherapy; reintroduced chemotherapy is considered only 1 line, e.g. platinum reintroduction in ovarian cancer). Exceptions must to be discussed with, and agreed by the Co-ordinating Investigator.
* Adequate hematological, liver and renal function, e.g.:
* Hemoglobin ≥9 mg/dl; Absolute Neutrophil Count (ANC) ≥1.5x109/l; platelets ≥100x109/l; normal coagulation factors (INR, PTT, PT).
* Serum bilirubin ≤upper normal limit (UNL); ALT, AST ≤ UNL but ≤ 2.5 x UNL in case of liver metastases; alkaline phosphatase (liver isoenzyme fraction) ≤ UNL or ≤1.5 x UNL of in case liver metastases; albumin within normal limits.
* Creatinine ≤1.5 mg/dl (≤133µmole/l) or calculated creatinine clearance ≥60 ml/min.
* Life expectancy of at least 3 months.
* Capability of understanding the nature of the trial and giving written informed consent.

Exclusion Criteria:

* Less than 4 weeks since last chemotherapy, radiotherapy or prior investigational therapy. Less than 2 weeks since last hormone or immunotherapy or signal transduction therapy.
* More than 30% liver parenchyma involvement assessed by computed tomography (CT) scan.
* History of hypersensitivity to preparations containing human albumin, and to intravenously administered proteins/peptides/antibodies.
* Active infection.
* Presence of cirrhosis with abnormal liver function test or chronic viral hepatitis.
* Presence of serious cardiac (congestive heart failure, angina pectoris, myocardial infarction within one year prior to study entry, uncontrolled hypertension or arrhythmia), neurological or psychiatric disorder.
* Presence of uncontrolled intercurrent illness or any condition which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study.
* Symptomatic brain metastases, primary brain tumors or leptomeningeal disease.
* Pregnancy or lactation, or unwillingness to use adequate method of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-02; Primary Completion 2008-11 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To determine of the maximum tolerated dose (MTD), based upon first cycle APO010-related DLT in patients with solid tumors. | 3 months

SECONDARY OUTCOMES:
A description of the frequency and severity of adverse events (AE) based on the NCI-CTC AE v.3.0. | 3 months
A description of the local toxicity at site of administration by route of administration based on the NCI-Common Terminology Criteria for Adverse Events (NCI-CTCAE v.3.0); the intervention required and by photographic record. | 3 months
A definition of the proportion of patients with neutralizing antibodies against APO010. | 3 months
A description of any objective tumor response based on modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Cristiana Sessa, Prof, MD, Principal Investigator — Oncology Institute of Southern Switzerland, Bellinzona Hospital, 6500 Bellinzona, Switzerland
Locations (2):
- Switzerland (2):
  - Oncology Institute of Southern Switzerland, Hospital of Bellinzona, Bellinzona
  - Multidisciplinary Oncology Center, Cantonal University Hospital of Vaud, Lausanne